CLINICAL TRIAL: NCT03451773
Title: A Phase IB/II Single-arm Study of M7824 (MSB0011359C) in Combination With Gemcitabine in Adults With Previously Treated Advanced Adenocarcinoma of the Pancreas
Brief Title: M7824 (MSB0011359C) in Combination With Gemcitabine in Adults With Previously Treated Advanced Adenocarcinoma of the Pancreas
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was closed after one treatment related death.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Udo Rudloff, MD, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 180061; 18-C-0061
Record Dates: First submitted 2018-03-01; First posted 2018-03-02 (Actual); Results first posted 2021-06-16 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-05

CONDITIONS: Cancer of Pancreas; Pancreas Cancer; Pancreatic Adenocarcinoma; Pancreatic Cancer; Pancreatic Neoplasms
Keywords: TGF Ligand Trap; Extracellular Domain of Human TGF Receptor II; Avelumab; Human IgG1 mAb Directed Against Human PD-L1; Health-Related Quality of Life
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/ Arm 1-Gemcitabine + de-escalating dose of M7824 (MSB0011359C) (Experimental): Gemcitabine (dose based on genetic testing results) + de-escalating dose of M7824
  Interventions: Drug: M7824; Drug: Gemcitabine
- 2/ Arm 2-Gemcitabine + Recommended Phase 2 Dose (RP2D) of M7824 (MSB0011359C) (Experimental): Gemcitabine (dose based on genetic testing results) + RP2D of M7824
  Interventions: Drug: M7824; Drug: Gemcitabine

INTERVENTIONS:
Drug: M7824 — 1,200 or 500mg every 2 weeks by intravenous (IV) infusion
  Other Names: MSB0011359C
Drug: Gemcitabine — Standard (1,000 mg/m^2) or reduced (600 mg/m^2 for 4 doses) intravenous (IV) once a week for first 4 weeks. Then, once weekly for 3 weeks with one week rest. Gemcitabine will be discontinued after 6 months of therapy
  Other Names: Gemzar

SUMMARY:
Background:

Pancreas cancer ranks 4th in all cancer-related deaths in the United States (U.S.) Gemcitabine is a standard treatment for it. M7824 (MSB0011359C) blocks a pathway that prevents the immune system from effectively fighting cancer. The two drugs together might help people with pancreas cancer.

Objective:

To test if giving M7824 together with gemcitabine is safe and causes tumors to shrink.

Eligibility:

People ages 18 and older with pancreatic cancer already treated with standard therapies

Design:

Participants will be screened with:

Medical history

Physical exam

Scans in a machine that takes pictures of the body

Blood, urine, and heart tests

Some participants may have a tumor sample removed.

Participants will get M7824 by intravenous (IV) once every 2 weeks. They will continue until their disease gets worse or they have unacceptable side effects.

After the first dose, participants will also get gemcitabine by IV once weekly for 7 weeks. Then they will get it as follows for up to 6 months: Skip 1 week, get the drug once a week for 3 weeks, skip 1 week.

Before treatment on the first day of each cycle, participants will repeat screening tests. They will also have:

Optional tumor biopsies before and after 3 cycles of therapy

Questions about their well-being and function

Genetic testing of tissue and blood samples

Participants will have a follow-up visit 4-5 weeks after they stop therapy. This includes a physical exam, blood and urine tests, and maybe a scan. If their disease does not get worse, they will be invited for scans every 12 weeks.

DETAILED DESCRIPTION:
Background:

* M7824 (MSB0011359C) is an investigational agent in phase IB/II clinical development with dual activity against transforming growth factor beta (TGF)-beta signaling (TGF-beta ligand trap; extracellular domain of human TGF-beta receptor II) and immune checkpoint ligand inhibition (PD-L1 inhibition; avelumab, fully human immunoglobulin G1 (IgG1) monoclonal antibody (mAb) directed against human PD-L1) with an acceptable toxicity profile and early signals of anti-cancer activity including in pancreas cancer.
* Gemcitabine (2 <=,2 <=-Difluorodeoxycytidine) is a standard-of-care nucleoside analogue in pancreas cancer with immunomodulatory mechanisms of actions in pancreas cancer patients.
* Preclinical studies in autochthonous and syngeneic murine models have shown that TGF-beta inhibition and PD-L1 inhibition cooperate with gemcitabine to achieve reduction of tumor growth and extension of survival induce anti-tumor immunity and reprogram the immune landscape.

Objectives:

* To determine the safety and tolerability of M7824 in combination with gemcitabine in subjects with metastatic or locally advanced pancreas cancer.
* To determine best overall response (BOR) rate according to Response Evaluation Criteria (Response Evaluation Criteria in Solid Tumors (RECIST) 1.1) in advanced pancreas cancer subjects.

Eligibility:

* Histologically confirmed diagnosis of adenocarcinoma of the pancreas.
* Patients must have progressed on prior chemotherapeutic regimen.
* Concurrent treatment with non-permitted drugs and other interventions, prior therapy with gemcitabine or any antibody / drug targeting T cell co-regulatory proteins (immune checkpoints) such as anti-PD 1, anti PD-L1, or anti-cytotoxic T lymphocyte antigen-4 (CTLA 4 antibody) is not allowed.

Design:

- The proposed study is a phase IB/II study of M7824 in combination with gemcitabine in a safety run-in of 6-18 patients and, if safe and tolerated, will proceed to an expansion phase II cohort with a standard Simon Minimax design.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patient must be able to understand and willing to sign a written informed consent document
* Age greater than of equal to 18 years. Because no dosing or adverse event data are currently available on the use of M7824 (MSB0011359C) in combination with gemcitabine in patients <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials
* Histologically or cytologically proven pancreatic adenocarcinoma (subjects with endocrine or acinar pancreatic carcinoma are not eligible).
* Patients must have disease that is not amenable to potentially curative resection.
* Subjects must have progressed on or after standard first-line systemic chemotherapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Must have evaluable or measurable disease per Response Evaluation in Solid Tumors (RECIST) 1.1.
* Adequate hematological function defined by:

  * white blood cell (WBC) count greater than or equal to 3x10(9)/L
  * with absolute neutrophil count (ANC) greater than or equal to 1.5x10(9)/L
  * lymphocyte count greater than or equal to 0.5x10(9)/L,
  * platelet count greater than or equal to 120x10(9)/L, and
  * Hemoglobin (Hgb) greater than or equal to 9 g/dL (in absence of blood transfusion)
* Adequate hepatic function defined by:

  * a total bilirubin level less than or equal to 1.5xUpper limit of normal (ULN),
  * an aspartate aminotransferase (AST) level less than or equal to 2.5xULN,
  * alanine aminotransferase (ALT) level less than or equal to 2.5Xuln.
* Adequate renal function defined by:

  * Creatinine up to 1.5 upper institutional limits OR creatinine clearance (CrCl) >50 mL/min/1.73 m^2 OR within normal as predicted by the Cockcroft-Gault formula:

Creatinine Clearance (CrCl)=(140-age) x (weight in kg) x (0.85, if female)/72 x Serum Creatinine (mg/dL)

- The effects of the study treatment on the developing human fetus are unknown; thus, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) within 28 days prior to study entry, for the duration of study participation and up to 120 days after the last dose of the drug. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

EXCLUSION CRITERIA:

* Patients who are receiving any other investigational agents
* Prior therapy with any antibody / drug targeting T cell coregulatory proteins (immune checkpoints) such as anti-Programmed cell death protein 1 (PD-1), anti-Programmed death-ligand 1 (PD-L1), or anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) antibody.
* Anticancer treatment within designated period before enrollment including:

  * minor surgical procedure (such as biliary stenting) within 14 days
  * major surgical procedure or radiation treatment within 28 days
  * chemotherapy or experimental drug treatment with published half-life known to be 72 hours within 14 days
  * experimental drug treatment with unpublished or half-life greater than 72 hours within 28 days
  * radiotherapy for measurable lesions delivered in a normal organ-sparing technique within 21 days (except for palliative radiotherapy)
* Concurrent treatment with non-permitted drugs including herbal remedies with immunostimulating properties (for example, mistletoe extract) or known to potentially interfere with major organ function (for example, hypericin).
* Previous malignant disease (other than the target malignancy to be investigated in this trial) within the last 3 years. Subjects with a history of cervical carcinoma in situ, superficial or no-invasive bladder cancer, or basal cell or squamous cell carcinoma in situ previously treated with curative intent are NOT excluded.
* Rapidly progressive disease which, in the opinion of the Investigator, may predispose to inability to tolerate treatment or trial procedures.
* Subjects with active central nervous system (CNS) metastases causing clinical symptoms or metastases that require therapeutic intervention are excluded. Subjects with a history of treated CNS metastases (by surgery or radiation therapy) are not eligible unless they have fully recovered from treatment, demonstrated no progression for at least 2 months, and do not require continued steroid therapy. Subjects with CNS metastases incidentally detected during Screening which do not cause clinical symptoms and for which standard of care suggests no therapeutic intervention is needed are eligible.
* Receipt of any organ transplantation, including allogeneic stem-cell transplantation, except of transplants that do not require immunosuppression (e.g., corneal transplant, hair transplant)
* Significant acute or chronic infections including tuberculosis (history of exposure or history of positive tuberculosis test; plus, presence of clinical symptoms, physical or radiographic findings)
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent with the exceptions:

  * diabetes type I, vitiligo, alopecia, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible;
  * subjects requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses less than or equal to 10 mg of prednisone or equivalent per day;
  * administration of steroids for other conditions through a route known to result in a minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation) is acceptable.
* Known severe hypersensitivity reactions to monoclonal antibodies (Grade greater than or equal to 3 National Cancer Institute Common Terminology Criteria in Adverse Events (NCI-CTCAE) v4.03, any history of anaphylaxis or history of uncontrolled asthma.
* Known severe hypersensitivity to gemcitabine.
* Female patients who are pregnant or breastfeeding. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with M7824 in combination with gemcitabine, breastfeeding should be discontinued.
* Known alcohol or drug abuse.
* Clinically significant cardiovascular / cerebrovascular disease as follows: cerebral vascular accident / stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (New York Heart Association Classification Class greater than or equal to II), or serious cardiac arrhythmia.
* Clinically relevant diseases (for example, inflammatory bowel disease) and/or uncontrolled medical conditions, which, in the opinion of the Investigator, might impair the subject's tolerance or ability to participate in the trial.
* Vaccine administration of live vaccines within 28 days of enrollment.
* Patients with known contrast allergies requiring pre-medication with steroids.
* Human immunodeficiency virus (HIV), hepatitis C virus (HCV), hepatitis B virus (HBV) positive patients on antiviral drugs are excluded due to the absence of previous experience with concurrent use of antiviral medications and the investigational drug product to be evaluated in the current study and possible for adverse pharmacokinetic and/or pharmacodynamic interactions.
* Known inherited bleeding disorder and/or history of bleeding diathesis such as von Willebrand factor (vWF) deficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2020-05-05 (Actual); Study Completion 2020-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Udo Rudloff, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Song S, Yuan P, Wu H, Chen J, Fu J, Li P, Lu J, Wei W. Dendritic cells with an increased PD-L1 by TGF-beta induce T cell anergy for the cytotoxicity of hepatocellular carcinoma cells. Int Immunopharmacol. 2014 May;20(1):117-23. doi: 10.1016/j.intimp.2014.02.027. Epub 2014 Mar 4. PMID 24606770
- [Background] Akhurst RJ, Hata A. Targeting the TGFbeta signalling pathway in disease. Nat Rev Drug Discov. 2012 Oct;11(10):790-811. doi: 10.1038/nrd3810. Epub 2012 Sep 24. PMID 23000686
- [Background] Ding X, Chen W, Fan H, Zhu B. Cytidine deaminase polymorphism predicts toxicity of gemcitabine-based chemotherapy. Gene. 2015 Mar 15;559(1):31-7. doi: 10.1016/j.gene.2015.01.010. Epub 2015 Jan 10. PMID 25582275
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-C-0061.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level -1: Gemcitabine + De-escalating Dose of M7824 (MSB0011359C): Gemcitabine (dose based on genetic testing results) + de-escalating dose of M7824
  M7824:500mg every 2 weeks by intravenous (IV) infusion
  Gemcitabine: Standard (1,000 mg/m^2) or reduced (600 mg/m^2 for 4 doses) intravenous (IV) once a week for first 4 weeks. Then, once weekly for 3 weeks with one week rest. Gemcitabine will be discontinued after 6 months of therapy
- Dose Level 0: Gemcitabine + Recommended Phase 2 Dose (RP2D) of M7824 (MSB0011359C): Gemcitabine (dose based on genetic testing results) + RP2D of M7824
  M7824: 1,200mg every 2 weeks by intravenous (IV) infusion
  Gemcitabine: Standard (1,000 mg/m^2) or reduced (600 mg/m^2 for 4 doses) intravenous (IV) once a week for first 4 weeks. Then, once weekly for 3 weeks with one week rest. Gemcitabine will be discontinued after 6 months of therapy
Period: Overall Study
Arm/Group | Dose Level -1: Gemcitabine + De-escalating Dose of M7824 (MSB0011359C) | Dose Level 0: Gemcitabine + Recommended Phase 2 Dose (RP2D) of M7824 (MSB0011359C)
Started | 1 | 6
Completed | 0 | 0
Not Completed | 1 | 6
Not completed — Death on study | 1 | 5
Not completed — Death during follow-up period | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level -1: Gemcitabine + De-escalating Dose of M7824 (MSB0011359C) | Dose Level 0: Gemcitabine + Recommended Phase 2 Dose (RP2D) of M7824 (MSB0011359C) | Total
Number analyzed (Participants) | 1 | 6 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 4 | 5
  >=65 years | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (0) | 55.87 (12.54) | 54.41 (12.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 0 | 4 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 1 | 5 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 5 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 | 6 | 7
Number of Participants with an Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1 [Count of Participants; unit: Participants] — ECOG is used by a clinician to describe a participant's level of functioning in activities of daily living. ECOG 0 is fully active. ECOG 1 is restricted in physically strenuous activity.
  Participants
    ECOG 0 | 1 | 3 | 4
    ECOG 1 | 0 | 3 | 3
Prior Therapy [Count of Participants; unit: Participants]
  Chemotherapy Multiple Agents Systemic | 1 | 6 | 7
  Surgery | 0 | 2 | 2
  Chemotherapy Single Agent Systemic | 0 | 3 | 3
  Limited Radiation | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Phase IB: Number and Severity of Grade 1-2 Adverse Events Possibly, Probably, or Definitely Related to Treatment
Description: Safety and tolerability of M7824 in combination with gemcitabine was assessed by the Common Terminology Criteria for Adverse Events (CTCAE)v5.0. Grade 1 is mild; asymptomatic or mild symptoms. Grade 2 is moderate; minimal non-invasive intervention indicated.
Time Frame: 30 days after treatment
Measure: Number; unit: adverse events
Arm/Group | Dose Level -1: Gemcitabine + De-escalating Dose of M7824 (MSB0011359C) | Dose Level 0: Gemcitabine + Recommended Phase 2 Dose (RP2D) of M7824 (MSB0011359C)
Number analyzed (Participants) | 1 | 6
adverse events
  Grade 1 Fatigue - Possibly Related | 1 | 2
  Grade 1 Vomiting - Possibly Related | 1 | 3
  Grade 1 Alanine aminotransferase increased - Possibly Related | 0 | 1
  Grade 1 Anemia - Possibly Related | 0 | 1
  Grade 1 Anorexia - Possibly Related | 0 | 1
  Grade 1 Aspartate aminotransferase increased - Possibly Related | 0 | 1
  Grade 1 Chills - Possibly Related | 0 | 2
  Grade 1 Dehydration - Possibly Related | 0 | 2
  Grade 1 Diarrhea - Possibly Related | 0 | 4
  Grade 1 Electrocardiogram QT corrected interval prolonged - Possibly Related | 0 | 1
  Grade 1 Fever - Possibly Related | 0 | 2
  Grade 1 Gastrointestinal disorders - Other, Gum bleeding - Possibly Related | 0 | 1
  Grade 1 Hyperglycemia - Possibly Related | 0 | 1
  Grade 1 Lymphocyte count decreased - Possibly Related | 0 | 1
  Grade 1 Nausea - Possibly Related | 0 | 1
  Grade 1 White blood cell decreased - Possibly Related | 0 | 1
  Grade 1 Bruising - Probably Related | 0 | 1
  Grade 1 Diarrhea - Probably Related | 1 | 1
  Grade 1 Lymphocyte count decreased - Probably Related | 0 | 1
  Grade 1 Platelet count decreased - Probably Related | 0 | 2
  Grade 1 Alanine aminotransferase increased - Definitely Related | 0 | 1
  Grade 2 Abdominal pain - Possibly Related | 0 | 1
  Grade 2 Alanine aminotransferase increased - Possibly Related | 0 | 1
  Grade 2 Anemia - Possibly Related | 0 | 1
  Grade 2 Aspartate aminotransferase increased - Possibly Related | 0 | 1
  Grade 2 Diarrhea - Possibly Related | 0 | 1
  Grade 2 Dyspnea - Possibly Related | 0 | 1
  Grade 2 Lymphocyte count decreased - Possibly Related | 0 | 3
  Grade 2 Nausea - Possibly Related | 0 | 1
  Grade 2 Neutrophil count decreased - Possibly Related | 0 | 4
  Grade 2 Platelet count decreased - Possibly Related | 0 | 1
  Grade 2 Tumor pain - Possibly Related | 0 | 1
  Grade 2 White blood cell decreased - Possibly Related | 0 | 2
  Grade 2 Anemia - Probably Related | 0 | 4
  Grade 2 Neutrophil count decreased - Probably Related | 0 | 1
  Grade 2 White blood cell decreased - Probably Related | 0 | 2
  Grade 2 Alkaline phosphatase increased - Definitely Related | 0 | 1
  Grade 2 Infusion related reaction - Definitely Related | 0 | 2

2. Primary Outcome: Phase IB: Number and Severity of Grade 3-5 Adverse Events Possibly, Probably, or Definitely Related to Treatment
Description: Safety and tolerability of M7824 in combination with gemcitabine was assessed by the Common Terminology Criteria for Adverse Events (CTCAE)v5.0. Grade 3 is severe or medically significant but not immediately life-threatening, Grade 4 is life-threatening consequences, and Grade 5 is death related to adverse event.
Time Frame: 30 days after treatment
Measure: Number; unit: adverse events
Arm/Group | Dose Level -1: Gemcitabine + De-escalating Dose of M7824 (MSB0011359C) | Dose Level 0: Gemcitabine + Recommended Phase 2 Dose (RP2D) of M7824 (MSB0011359C)
Number analyzed (Participants) | 1 | 6
adverse events
  Grade 3 Anemia - Possibly Related | 0 | 1
  Grade 3 Diarrhea Possibly Related | 0 | 2
  Grade 3 Nausea - Possibly Related | 0 | 1
  Grade 3 Neutrophil count decreased - Possibly Related | 0 | 1
  Grade 3 Platelet Count Decreased - Possibly Related | 0 | 1
  Grade 3 Pleural Effusion - Possibly Related | 0 | 1
  Grade 3 Anemia Probably Related | 0 | 1
  Grade 3 Lymphocyte Count Decreased - Probably Related | 0 | 1
  Grade 3 Platelet Count Decreased - Probably Related | 0 | 2
  Grade 3 White Blood Cell Decreased - Probably Related | 0 | 1
  Grade 3 Alanine Aminotransferase Increased - Definitely Related | 0 | 1
  Grade 3 Lipase Increased - Definitely Related | 0 | 1
  Grade 4 Neutrophil count decreased - Probably Related | 0 | 1
  Grade 4 Aspartate Aminotransferase increased - Definitely Related | 0 | 1
  Grade 5 Immune Checkpoint Inhibitor (ICI)-Induced Hepatitis - Definitely Related | 0 | 1

3. Primary Outcome: Phase II: Number of Participants With a Best Overall Response (BOR)
Description: Changes in tumor size and occurrence of metastases was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1 to determine the best overall response: Complete Response (CR), Partial Response (PR), and Stable Disease (SD), whichever is recorded first. Complete Response is disappearance of all lesions, Partial Response is at least a 30% decrease in the sum of diameters of target lesions, and Stable Disease is when the sum of all target lesions does not qualify for CR, PR, or Progressive Disease (PD), defined as the appearance of new lesions.
Time Frame: Every 8 weeks, up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level -1: Gemcitabine + De-escalating Dose of M7824 (MSB0011359C) | Dose Level 0: Gemcitabine + Recommended Phase 2 Dose (RP2D) of M7824 (MSB0011359C)
Number analyzed (Participants) | 1 | 6
Participants
  Complete Response | 0 | 0
  Partial Response | 0 | 0
  Stable Disease | 1 | 3
  Progressive Disease | 0 | 0

4. Primary Outcome: Duration of Treatment-related Adverse Events (AEs)
Description: Duration of treatment-related AE's is defined as the time from the date treatment consent signed to end of treatment. Grade 1-4 adverse events observed in participants with pancreatic cancer assessed by the Common Terminology Criteria in Adverse Events (CTCAE) v5.0. Grade 1 is mild. Grade 2 is moderate. Grade 3 is severe or medically significant. And Grade 4 is life-threatening.
Time Frame: Time to resolution of adverse events, which is the time recorded until it took for the adverse event to resolve to grade 1 or less (if there is a death, it is that time), approximately 12 months.
Population: * = death. Zero = adverse event started and resolved on the same day and/or participant died.
Measure: Number; unit: Days
Arm/Group | Dose Level -1: Gemcitabine + De-escalating Dose of M7824 (MSB0011359C) | Dose Level 0: Gemcitabine + Recommended Phase 2 Dose (RP2D) of M7824 (MSB0011359C)
Number analyzed (Participants) | 1 | 6
Days
  Pt 6 - Grade 1 Diarrhea: number analyzed (Participants) | 1 | 0
  Pt 6 - Grade 1 Diarrhea | 45 |
  Pt 6 - Grade 1 Fatigue: number analyzed (Participants) | 1 | 0
  Pt 6 - Grade 1 Fatigue | 0 |
  Pt 6 - Grade 1 Vomiting: number analyzed (Participants) | 1 | 0
  Pt 6 - Grade 1 Vomiting | 0 |
  Pt 1 - Grade 1 Alanine aminotransferase increased: number analyzed (Participants) | 0 | 1
  Pt 1 - Grade 1 Alanine aminotransferase increased |  | 172
  Pt 7 - Grade 1 Alanine aminotransferase increased: number analyzed (Participants) | 0 | 1
  Pt 7 - Grade 1 Alanine aminotransferase increased |  | 1
  Pt 2 - Grade 1 Anemia: number analyzed (Participants) | 0 | 1
  Pt 2 - Grade 1 Anemia |  | 1
  Pt 4* - Grade 1 Anorexia: number analyzed (Participants) | 0 | 1
  Pt 4* - Grade 1 Anorexia |  | 27
  Pt 1* - Grade 1 Aspartate aminotransferase increased: number analyzed (Participants) | 0 | 1
  Pt 1* - Grade 1 Aspartate aminotransferase increased |  | 173
  Pt 5* - Grade 1 Bruising: number analyzed (Participants) | 0 | 1
  Pt 5* - Grade 1 Bruising |  | 17
  Pt 5 - Grade 1 Chills first occurrence: number analyzed (Participants) | 0 | 1
  Pt 5 - Grade 1 Chills first occurrence |  | 0
  Pt 5 - Grade 1 Chills second occurrence: number analyzed (Participants) | 0 | 1
  Pt 5 - Grade 1 Chills second occurrence |  | 0
  Pt 1 - Grade Dehydration: number analyzed (Participants) | 0 | 1
  Pt 1 - Grade Dehydration |  | 2
  Pt 2* - Dehydration: number analyzed (Participants) | 0 | 1
  Pt 2* - Dehydration |  | 301
  Pt 1 - Grade 1 Diarrhea: number analyzed (Participants) | 0 | 1
  Pt 1 - Grade 1 Diarrhea |  | 3
  Pt 2 - Grade 1 Diarrhea first occurrence: number analyzed (Participants) | 0 | 1
  Pt 2 - Grade 1 Diarrhea first occurrence |  | 4
  Pt 2 - Grade 1 Diarrhea second occurrence: number analyzed (Participants) | 0 | 1
  Pt 2 - Grade 1 Diarrhea second occurrence |  | 19
  Pt 5 - Grade 1 Diarrhea: number analyzed (Participants) | 0 | 1
  Pt 5 - Grade 1 Diarrhea |  | 0
  Pt 5* - Grade 1 Electrocardiogram QT corrected interval prolonged: number analyzed (Participants) | 0 | 1
  Pt 5* - Grade 1 Electrocardiogram QT corrected interval prolonged |  | 31
  Pt 1 - Grade 1 Fatigue: number analyzed (Participants) | 0 | 1
  Pt 1 - Grade 1 Fatigue |  | 2
  Pt 2* - Grade 1 Fatigue: number analyzed (Participants) | 0 | 1
  Pt 2* - Grade 1 Fatigue |  | 330
  Pt 1 - Grade 1 Fever: number analyzed (Participants) | 0 | 1
  Pt 1 - Grade 1 Fever |  | 4
  Pt 5 - Grade 1 Fever: number analyzed (Participants) | 0 | 1
  Pt 5 - Grade 1 Fever |  | 0
  Pt 3 - Grade 1 Gastrointestinal disorder - Other, specify: number analyzed (Participants) | 0 | 1
  Pt 3 - Grade 1 Gastrointestinal disorder - Other, specify |  | 56
  Pt 1* - Grade 1 Hyperglycemia: number analyzed (Participants) | 0 | 1
  Pt 1* - Grade 1 Hyperglycemia |  | 151
  Pt 2 - Grade 1 Lymphocyte count decreased first occurrence: number analyzed (Participants) | 0 | 1
  Pt 2 - Grade 1 Lymphocyte count decreased first occurrence |  | 16
  Pt 2 - Lymphocyte count decreased second occurrence: number analyzed (Participants) | 0 | 1
  Pt 2 - Lymphocyte count decreased second occurrence |  | 5
  Pt 5 - Grade 1 Nausea: number analyzed (Participants) | 0 | 1
  Pt 5 - Grade 1 Nausea |  | 0
  Pt 2 - Grade 1 Platelet count decreased: number analyzed (Participants) | 0 | 1
  Pt 2 - Grade 1 Platelet count decreased |  | 14
  Pt 3* - Grade 1 Platelet count decreased: number analyzed (Participants) | 0 | 1
  Pt 3* - Grade 1 Platelet count decreased |  | 50
  Pt 1 - Grade 1 Vomiting: number analyzed (Participants) | 0 | 1
  Pt 1 - Grade 1 Vomiting |  | 3
  Pt 5 - Grade 1 Vomiting: number analyzed (Participants) | 0 | 1
  Pt 5 - Grade 1 Vomiting |  | 0
  Pt 7* - Grade 1 Vomiting: number analyzed (Participants) | 0 | 1
  Pt 7* - Grade 1 Vomiting |  | 1
  Pt 2 - Grade 1 White blood cell decreased: number analyzed (Participants) | 0 | 1
  Pt 2 - Grade 1 White blood cell decreased |  | 327
  Pt 1* - Grade 2 Abdominal pain: number analyzed (Participants) | 0 | 1
  Pt 1* - Grade 2 Abdominal pain |  | 167
  Pt 1 - Grade 2 Alanine aminotransferase increased: number analyzed (Participants) | 0 | 1
  Pt 1 - Grade 2 Alanine aminotransferase increased |  | 1
  Pt 7* - Grade 2 Alkaline aminotransferase increased: number analyzed (Participants) | 0 | 1
  Pt 7* - Grade 2 Alkaline aminotransferase increased |  | 0
  Pt 2 - Grade 2 Anemia: number analyzed (Participants) | 0 | 1
  Pt 2 - Grade 2 Anemia |  | 14
  Pt 5 - Grade 2 Anemia first occurrence: number analyzed (Participants) | 0 | 1
  Pt 5 - Grade 2 Anemia first occurrence |  | 1
  Pt 5 - Grade 2 Anemia second occurrence: number analyzed (Participants) | 0 | 1
  Pt 5 - Grade 2 Anemia second occurrence |  | 5
  Pt 3 - Grade 2 Anemia: number analyzed (Participants) | 0 | 1
  Pt 3 - Grade 2 Anemia |  | 14
  Pt 2* - Grade 2 Anemia: number analyzed (Participants) | 0 | 1
  Pt 2* - Grade 2 Anemia |  | 327
  Pt 3 - Grade 2 Aspartate aminotransferase increased: number analyzed (Participants) | 0 | 1
  Pt 3 - Grade 2 Aspartate aminotransferase increased |  | 1
  Pt 2 - Grade 2 Diarrhea: number analyzed (Participants) | 0 | 1
  Pt 2 - Grade 2 Diarrhea |  | 10
  Pt 1* - Grade 2 Dyspnea: number analyzed (Participants) | 0 | 1
  Pt 1* - Grade 2 Dyspnea |  | 176
  Pt 1 - Grade 1 Infusion related reaction first occurrence: number analyzed (Participants) | 0 | 1
  Pt 1 - Grade 1 Infusion related reaction first occurrence |  | 0
  Pt 1 - Grade 2 Infusion related reaction second occurrence: number analyzed (Participants) | 0 | 1
  Pt 1 - Grade 2 Infusion related reaction second occurrence |  | 0
  Pt 2* - Grade 2 Lymphocyte count decreased: number analyzed (Participants) | 0 | 1
  Pt 2* - Grade 2 Lymphocyte count decreased |  | 322
  Pt 3 - Grade 2 Lymphocyte count decreased first occurrence: number analyzed (Participants) | 0 | 1
  Pt 3 - Grade 2 Lymphocyte count decreased first occurrence |  | 1
  Pt 3* - Grade 2 Lymphocyte count decreased second occurrence: number analyzed (Participants) | 0 | 1
  Pt 3* - Grade 2 Lymphocyte count decreased second occurrence |  | 32
  Pt 7 - Grade 2 Nausea: number analyzed (Participants) | 0 | 1
  Pt 7 - Grade 2 Nausea |  | 1
  Pt 2 - Grade 2 Neutrophil count decreased: number analyzed (Participants) | 0 | 1
  Pt 2 - Grade 2 Neutrophil count decreased |  | 2
  Pt 3 - Grade 2 Neutrophil count decreased first occurrence: number analyzed (Participants) | 0 | 1
  Pt 3 - Grade 2 Neutrophil count decreased first occurrence |  | 14
  Pt 3 - Grade 2 Neutrophil count decreased second occurrence: number analyzed (Participants) | 0 | 1
  Pt 3 - Grade 2 Neutrophil count decreased second occurrence |  | 1
  Pt 3 - Grade 2 Neutrophil count decreased third occurrence: number analyzed (Participants) | 0 | 1
  Pt 3 - Grade 2 Neutrophil count decreased third occurrence |  | 1
  Pt 2* - Grade 2 Neutrophil count decreased: number analyzed (Participants) | 0 | 1
  Pt 2* - Grade 2 Neutrophil count decreased |  | 327
  Pt 2* - Grade 2 Platelet count decreased: number analyzed (Participants) | 0 | 1
  Pt 2* - Grade 2 Platelet count decreased |  | 327
  Pt 7* - Grade 2 Tumor pain: number analyzed (Participants) | 0 | 1
  Pt 7* - Grade 2 Tumor pain |  | 11
  Pt 2 - Grade White blood cell decreased: number analyzed (Participants) | 0 | 1
  Pt 2 - Grade White blood cell decreased |  | 2
  Pt 3 - Grade 2 White blood cell decreased first occurrence: number analyzed (Participants) | 0 | 1
  Pt 3 - Grade 2 White blood cell decreased first occurrence |  | 0
  Pt 3 - Grade 2 White blood cell decreased second occurrence: number analyzed (Participants) | 0 | 1
  Pt 3 - Grade 2 White blood cell decreased second occurrence |  | 0
  Pt 3 - Grade 2 White blood cell decreased third occurrence: number analyzed (Participants) | 0 | 1
  Pt 3 - Grade 2 White blood cell decreased third occurrence |  | 0
  Pt 7* - Grade 3 Alanine aminotransferase increased: number analyzed (Participants) | 0 | 1
  Pt 7* - Grade 3 Alanine aminotransferase increased |  | 0
  Pt 2* - Grade 3 Anemia: number analyzed (Participants) | 0 | 1
  Pt 2* - Grade 3 Anemia |  | 2
  Pt 5 - Grade 3 Anemia: number analyzed (Participants) | 0 | 1
  Pt 5 - Grade 3 Anemia |  | 1
  Pt 2 - Grade 3 Diarrhea first occurrence: number analyzed (Participants) | 0 | 1
  Pt 2 - Grade 3 Diarrhea first occurrence |  | 0
  Pt 2 - Grade 3 Diarrhea second occurrence: number analyzed (Participants) | 0 | 1
  Pt 2 - Grade 3 Diarrhea second occurrence |  | 6
  Pt 7* - Grade 3 Lipase increased: number analyzed (Participants) | 0 | 1
  Pt 7* - Grade 3 Lipase increased |  | 1
  Pt 3 - Grade 3 Lymphocyte count decreased: number analyzed (Participants) | 0 | 1
  Pt 3 - Grade 3 Lymphocyte count decreased |  | 1
  Pt 7* - Grade 3 Nausea: number analyzed (Participants) | 0 | 1
  Pt 7* - Grade 3 Nausea |  | 1
  Pt 3 - Grade 3 Neutrophil count decreased: number analyzed (Participants) | 0 | 1
  Pt 3 - Grade 3 Neutrophil count decreased |  | 0
  Pt 2 - Grade 3 Platelet count decreased: number analyzed (Participants) | 0 | 1
  Pt 2 - Grade 3 Platelet count decreased |  | 3
  Pt 5 - Grade 3 Platelet count decreased first occurrence: number analyzed (Participants) | 0 | 1
  Pt 5 - Grade 3 Platelet count decreased first occurrence |  | 2
  Pt 5 - Grade 3 Platelet count decreased second occurrence: number analyzed (Participants) | 0 | 1
  Pt 5 - Grade 3 Platelet count decreased second occurrence |  | 5
  Pt 3 - Grade 3 Pleural effusion: number analyzed (Participants) | 0 | 1
  Pt 3 - Grade 3 Pleural effusion |  | 8
  Pt 3 - Grade 3 White blood cell decreased: number analyzed (Participants) | 0 | 1
  Pt 3 - Grade 3 White blood cell decreased |  | 14
  Pt 7* - Grade 4 Aspartate aminotransferase increased: number analyzed (Participants) | 0 | 1
  Pt 7* - Grade 4 Aspartate aminotransferase increased |  | 1
  Pt 3 - Grade 4 Neutrophil count decreased: number analyzed (Participants) | 0 | 1
  Pt 3 - Grade 4 Neutrophil count decreased |  | 14
  Pt 7 - Grade 5 Immune system disorders - Other, Specify: number analyzed (Participants) | 0 | 1
  Pt 7 - Grade 5 Immune system disorders - Other, Specify |  | 0

5. Secondary Outcome: Number of Participants With an Immune-related Best Overall Response (irBOR)
Description: irBOR is defined as the duration of immune-related best overall response measured from the time measurement criteria are met for Immune-related Complete Response (irCR) or Immune-related Partial Response (irPR) (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented. Immune related changes in tumor size and occurrence of metastases was assessed by the Modified Immune-related Response Evaluation Criteria in Solid Tumors (irRECIST). Immune-related Complete Response (irCR) is complete disappearance of all lesions and no new lesions. Immune-related Partial Response (irPR) is sum of the longest diameters of target and new measurable lesions neither irCR, irPR (compared to baseline) or irPD (compared to nadir). Immune-related Progressive Disease (irPD) is appearance of new lesions.
Time Frame: Every 6-12 weeks, up to 1 year
Population: This outcome measure was not done because no participants lived long enough to have confirmatory scans to confirm immune related response.
Arm/Group | Dose Level -1: Gemcitabine + De-escalating Dose of M7824 (MSB0011359C) | Dose Level 0: Gemcitabine + Recommended Phase 2 Dose (RP2D) of M7824 (MSB0011359C)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Percentage of Evaluable Participants Alive at 6 Months and 9 Months
Description: Participants who are alive at 6 months and 9 months after therapy.
Time Frame: At 6 and 9 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Level -1: Gemcitabine + De-escalating Dose of M7824 (MSB0011359C) | Dose Level 0: Gemcitabine + Recommended Phase 2 Dose (RP2D) of M7824 (MSB0011359C)
Number analyzed (Participants) | 1 | 6
percentage of participants
  6 Months | NA [NA to NA] — Since only one participant was accrued to this cohort, no median survival times can be given. The participant progressed and died. | 33.3 [4.6 to 62.6]
  9 Months | NA [NA to NA] — Since only one participant was accrued to this cohort, no median survival times can be given. The participant progressed and died. | 16.7 [0.8 to 51.7]

7. Secondary Outcome: Percentage of Participants Who Have Not Progressed at 3 Months
Description: Percentage of participants who have not progressed at 3 months. Progression was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) and is defined as the appearance of new lesions.
Time Frame: 3 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Level -1: Gemcitabine + De-escalating Dose of M7824 (MSB0011359C) | Dose Level 0: Gemcitabine + Recommended Phase 2 Dose (RP2D) of M7824 (MSB0011359C)
Number analyzed (Participants) | 1 | 6
percentage of participants | NA [NA to NA] — Since only one participant was accrued to this cohort, no median survival times can be given. The participant progressed and died. | 16.7 [0.8 to 51.7]

8. Secondary Outcome: Overall Median Survival
Description: OS is the median amount of time subject survives after therapy.
Time Frame: up to 1 year
Population: On participant died.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- All Participants: All participants in Dose Level -1: Gemcitabine + De-escalating Dose of M7824 (MSB0011359C), and Dose Level 0: Gemcitabine + Recommended Phase 2 Dose (RP2D) of M7824 (MSB0011359C)
Arm/Group | All Participants
Number analyzed (Participants) | 6
Months | 3.5 [0.5 to 11.7]

9. Secondary Outcome: Overall Progression Free Survival
Description: PFS is the median amount of time subject survives without disease progression after treatment. Progression was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) and is defined as the appearance of new lesions.
Time Frame: up to 6 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | All Participants
Number analyzed (Participants) | 7
Months | 1.4 [0.5 to 5.1]

10. Other Pre Specified Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 7 months and 20 days for Dose Level -1, and 15 months and 20 days for Dose Level 0.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level -1: Gemcitabine + De-escalating Dose of M7824 (MSB0011359C) | Dose Level 0: Gemcitabine + Recommended Phase 2 Dose (RP2D) of M7824 (MSB0011359C)
Number analyzed (Participants) | 1 | 6
Participants | 1 | 6

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 7 months and 20 days for Dose Level -1, and 15 months and 20 days for Dose Level 0.
Arm/Group | Dose Level -1: Gemcitabine + De-escalating Dose of M7824 (MSB0011359C) | Dose Level 0: Gemcitabine + Recommended Phase 2 Dose (RP2D) of M7824 (MSB0011359C)
All-Cause Mortality (participants affected / at risk) | 1/1 | 6/6
Serious Adverse Events (participants affected / at risk) | 0/1 | 6/6
Other Adverse Events (participants affected / at risk) | 1/1 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level -1: Gemcitabine + De-escalating Dose of M7824 (MSB0011359C) (N=1) | Dose Level 0: Gemcitabine + Recommended Phase 2 Dose (RP2D) of M7824 (MSB0011359C) (N=6)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 4 (5)
Disease progression (General disorders) | 0 (0) | 2 (2)
Duodenal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Immune system disorders - Other, Immune checkpoint inhibitor (ICI)- induced hepatitis (Immune system disorders) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level -1: Gemcitabine + De-escalating Dose of M7824 (MSB0011359C) (N=1) | Dose Level 0: Gemcitabine + Recommended Phase 2 Dose (RP2D) of M7824 (MSB0011359C) (N=6)
Abdominal pain (Gastrointestinal disorders) | 1 (3) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 4 (9)
Fatigue (General disorders) | 1 (1) | 3 (3)
Gastrointestinal disorders - Other, Abdominal cramp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, pale bowel movement (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, Gum bleeding (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastrointestinal disorders - Other, Malena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Angular chelitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Granular irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (6)
Weight loss (Investigations) | 1 (2) | 1 (5)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (4)
Alkaline phosphatase increased (Investigations) | 0 (0) | 4 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 4 (9)
Ascites (Gastrointestinal disorders) | 0 (0) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 4 (4)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Bloating (Gastrointestinal disorders) | 0 (0) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (2)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Gastrointestinal disorders) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 1 (3)
Dysarthria (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (5)
Ear and labyrinth disorders - Other, Right ear swelling (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 1 (2)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 2 (2)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (6)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (7)
Pancreatic enyzme decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 4 (7)
Weight gain (Investigations) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 2 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Dysarthia (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-20): https://cdn.clinicaltrials.gov/large-docs/73/NCT03451773/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-18): https://cdn.clinicaltrials.gov/large-docs/73/NCT03451773/ICF_001.pdf